CLINICAL TRIAL: NCT03185221
Title: Comparing the Safety and Efficacy of Cordimax and Xience V Drug-eluting Stents, for the Treatment of Coronary Heart Disease (CHD) in the Clinical Research of Real World
Brief Title: Cordimax China Post Market Surveillance
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shandong Branden Med.Device Co.,Ltd (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Branden-456
Record Dates: First submitted 2017-05-16; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Coronary Artery Stenosis
Keywords: Stents Coronary Artery Disease
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cordimax (Experimental): Rapamycin Eluting Coronary Stent
  Interventions: Device: Cordimax
- XIENCE V (Active Comparator): Everolimus Eluting Coronary Stent
  Interventions: Device: XIENCE V

INTERVENTIONS:
Device: Cordimax — One rapamycin eluting stent for treating the adapted coronary patients
  Arms: Cordimax
Device: XIENCE V — One everolimus eluting stent for treating the adapted coronary patients
  Arms: XIENCE V

SUMMARY:
Study purpose: This study is a prospective, randomized, controlled multicenter clinical research, which is to assess the effect of Cordimax and Xience V drug-eluting stents as they dealing with all kinds of complex lesions in the real world.

Study group Experimental group: Cordimax® Rapamycin Eluting Coronary Stent System Control group: XIENCE V® Everolimus Eluting Coronary Stent System

DETAILED DESCRIPTION:
The purpose of the post market clinical trial is to evaluate the safety and efficacy of the Cordimax Rapamycin Eluting Coronary Stent System (RECS). The Cordimax will be compared to an active control group represented by the FDA approved commercially available Abbott Vascular XIENCE V® EECS Everolimus Eluting Coronary Stent System.

The post market clinical trial consists of a randomized clinical trial (RCT) in China which will enroll approximately 3660 subjects (2:1 randomization Cordimax® RECS : XIENCE V® EECS) with a maximum of two de novo native coronary artery lesion treatment within vessel sizes >= 2.5 mm and <= 4 mm.

All subjects in the RCT will be screened per the protocol required inclusion/exclusion criteria. The data collected will be compared to data from the subjects enrolled into the XIENCE V® arm of US RCT.

All subjects will have clinical follow-up at 30, 60, 90days, and 1, 2, 3, 4, and 5 years so as to collect the needed data for the subsequent analysis.(Data collecting at 1st year will be conducted in the clinic in order to get the 12 lead ecg result once after out of the hospital) .

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years old or more
2. patients with symptomatic coronary artery disease
3. adapt to the DES treatment according to guide
4. with one or more in diameter of the stenosis of 50% or more coronary artery lesions (refer to 2.5~4.0 mm) in diameter ;has the objective basis of myocardial ischemia
5. patients willing to participate and sign in research

Exclusion Criteria:

1. Women in pregnancy or lactation
2. Patients are not adapt to the antiplatelet and/or anticoagulant therapy in the expectation
3. Patients were banned to use the antiplatelet and/or anticoagulant therapy
4. Patients have participated in other devices or drugs or other research at the same time, and have not yet reached the end of the research project
5. Patients who must stop clopidogrel to accept a elective surgery
6. patients that the researchers think who are not suitable for stent placement and unable to complete the follow-up, such as the late malignant tumor patients, patients with severe liver and kidney disease, cerebral apoplexy patients, severe infection and severe patients with diseases of the blood system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3660 (Actual)
Dates: Start 2013-06-20 (Actual); Primary Completion 2019-06-20 (Estimated); Study Completion 2020-06-20 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure(TLF) | at 1st year
  including Cardiac death, target vessel myocardial infarction, and clinical symptom driven target vessel revascularization

SECONDARY OUTCOMES:
Thrombotic events incidence | at30 60 90 days and 1st 2st 3st 4st 5st year
  According to ARC definition it includes deterministic thrombosis, possible thrombosis and not eliminating thrombosis; point-in-time include acute within 24h, subacute between 2 and 30 d and later period over 30 d
Major adverse cardiovascular events (MACE) | at30 60 90 days and 1st 2st 3st 4st 5st year
  Events include cardiac death, myocardial infarction of target vessel and target lesion revascularization (TLR) by clinical-driven
The Success Rate of Stent Placement | in the operation
  The stent can arrive and through the target lesion area, and can be expanded finally.
Operation Success Rate | 0 to 24 hours after intervention
  After stent implantation, stent diameter stenosis < 30% (visual), TIMI flow class 3, and hospitalization MACE events did not happen.
Cost of the hospitalization | 0 to 24hours after discharge
  The total expenses in the process of operation
Length of stay | 0 to 24 hours after discharge
  The total time consumption in the process of operation

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No